CLINICAL TRIAL: NCT05088356
Title: Phase 1 Trial for Patients With Advanced Hematologic Malignancies Undergoing Reduced Intensity Allogeneic HCT With a T-cell Depleted Graft With Infusion of Conventional T-cells and Regulatory T-cells
Brief Title: Reduced Intensity Allogeneic HCT in Advanced Hematologic Malignancies w/T-Cell Depleted Graft
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-60439; BMT372 (Other: Stanford); NCI-2021-12228 (Other: NCI Trial ID)
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation (HCT); Advanced Hematologic Malignancies; Acute Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders
Keywords: Reduced intensity conditioning (RIC); GVHD
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — fludarabine; fludarabine phosphate; Melphalan; Tacrolimus; Cyclophosphamide; Alkylating Agents; plerixafor; Granulocyte Colony-Stimulating Factor; Thiotepa; Mycophenolic Acid; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Arm A1: Matched related/matched unrelated donor transplantation (closed) (Experimental): Subjects will receive reduced intensity preparative chemotherapy conditioning for a matched related/ unrelated donor transplant:.
  * Fludarabine (160 mg/m2)
  * Melphalan (50 mg/m2)
  * TBI (4Gy)
  All enrolled subjects will receive GVHD prophylaxis with single-agent tacrolimus.
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Melphalan; Drug: Tacrolimus; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent
- Arm B: Haploidentical transplantation (closed) (Experimental): Subjects without an identified matched related or matched unrelated donor will receive a haploidentical transplantation with reduced intensity preparative conditioning:
  -. Fludarabine (160 mg/m2)
  * Melphalan (100 mg/m2
  * TBI (4Gy)
  Patients will receive GVHD prophylaxis with post-transplant cyclophosphamide and tacrolimus.
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Melphalan; Device: CliniMACS CD34 Reagent System; Drug: Tacrolimus; Drug: Cyclophosphamide; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent
- Arm A2: Fully matched (8/8) related/unrelated donor transplantation (Experimental): Subjects will receive reduced intensity preparative chemotherapy conditioning for a matched related/ unrelated donor transplant:
  * Fludarabine (160 mg/m2)
  * Thiotepa (10 mg/kg)
  * TBI (4Gy)
  All enrolled subjects will receive GVHD prophylaxis with single-agent tacrolimus.
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Tacrolimus; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent; Drug: Thiotepa
- Arm A3: Fully (8/8) matched related/unrelated donor transplantation (Experimental): Subjects will receive reduced intensity preparative chemotherapy conditioning for a matched related/ unrelated donor transplant:
  * Fludarabine (160 mg/m2)
  * Thiotepa (5 mg/kg)
  * TBI (2-3 Gy).
  All enrolled subjects will receive GVHD prophylaxis with single-agent tacrolimus.
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Tacrolimus; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent; Drug: Thiotepa
- Arm C1:7/8 mismatched related/unrelated donor transplantation (closed) (Experimental): Subjects will receive reduced intensity preparative chemotherapy conditioning for a matched related/ unrelated donor transplant:
  * Fludarabine (160 mg/m2)
  * Thiotepa (10 mg/kg)
  * TBI (4 Gy) All enrolled subjects will receive GVHD prophylaxis with tacrolimus and mycophenolate mofetil (MMF).
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Tacrolimus; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent; Drug: Thiotepa; Drug: Mycophenolate Mofetil (MMF)
- Arm C2: 7/8 mismatched related/unrelated donor transplantation (Experimental): Subjects will receive reduced intensity preparative chemotherapy conditioning for a matched related/ unrelated donor transplant:
  * Fludarabine (160 mg/m2)
  * Thiotepa (5 mg/kg)
  * TBI (2-3 Gy)
  All enrolled subjects will receive GVHD prophylaxis with tacrolimus and ruxolitinib.
  Interventions: Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC; Drug: Fludarabine; Drug: Tacrolimus; Drug: Plerixafor; Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent; Drug: Thiotepa; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Purified regulatory T-cells (Treg) plus CD34+ HSPC — Purified regulatory T-cells (Treg) plus CD34+ hematopoietic progenitor cells ("CD34+ HSPC"), followed by conventional T-cells (Tcon) Manufactured at SCTT Laboratory, dose 1x10^6 cells/ kg to 3x10^6 cells/kg
Drug: Fludarabine — Fludarabine (160 mg/m2)
  Other Names: Beneflur; SH T 586; fludarabine monophosphate
Drug: Melphalan — Melphalan (50 mg/m2)
  Other Names: Melphalanum
  Arms: Arm A1: Matched related/matched unrelated donor transplantation (closed); Arm B: Haploidentical transplantation (closed)
Device: CliniMACS CD34 Reagent System — The CliniMACS® CD34 Reagent System is a medical device that is used in vitro to select and enrich specific cell populations is manufactured by Miltenyi Biotec
  Arms: Arm B: Haploidentical transplantation (closed)
Drug: Tacrolimus — 4-6ng/mL
  Other Names: Prograf; Advagraf; fujimycin
Drug: Cyclophosphamide — 40mg/kg
  Other Names: alkylating agent
  Arms: Arm B: Haploidentical transplantation (closed)
Drug: Plerixafor — Dose 0.24 mg/kg, manufactured by Genzyme
  Other Names: Mozobil; AMD 3100; LM-3100
Drug: Filgrastim granulocyte colony-stimulating factor (G-CSF) or equivalent — Single-use vials contain either 300 mcg or 480 mcg filgrastim at a fill volume of 1.0 mL or 1.6 mL
  Other Names: filgrastim XM02
Drug: Thiotepa — Thiotepa 10 mg/kg
  Other Names: Tepandina
  Arms: Arm A2: Fully matched (8/8) related/unrelated donor transplantation; Arm A3: Fully (8/8) matched related/unrelated donor transplantation; Arm C1:7/8 mismatched related/unrelated donor transplantation (closed); Arm C2: 7/8 mismatched related/unrelated donor transplantation
Drug: Mycophenolate Mofetil (MMF) — MMF 1000 mg BID
  Other Names: CellCept
  Arms: Arm C1:7/8 mismatched related/unrelated donor transplantation (closed)
Drug: Ruxolitinib — Ruxolitinib 5 mg BID
  Other Names: Jakafi
  Arms: Arm C2: 7/8 mismatched related/unrelated donor transplantation

SUMMARY:
Reduced intensity conditioning (RIC) has emerged and been increasingly adopted as a modality to allow preparative conditioning pre transplant to be tolerated by older adults or those patients that are otherwise unfit for myeloablative conditioning. In this study, we aim to use RIC followed by matched related/unrelated donor, 7/8 matched related/unrelated donor, or haploidentical donor peripheral blood stem cell transplantation. Standard strategies to control the alloreactivity following HCT utilize immunosuppressive or cytotoxic medications. In this study, we explore donor graft engineering to enrich for immmunoregulatory populations to facilitate post transplantation immune reconstitution while minimizing graft versus host disease (GVHD) with post-transplant immunosuppressive agents.

DETAILED DESCRIPTION:
The objectives for the study are listed below:

Primary Objectives

*Determine the safety, and feasibility of administration of several dose combinations of conventional T-cells (Tcon) and regulatory T-cells (Treg) in subjects undergoing allogeneic hematopoietic cell transplantation (HCT) with related/unrelated HLA-matched or mismatched donors, or haploidentical donors with reduced intensity conditioning preparative regimen.

Secondary Objectives

* To determine the GVHD-free relapse-free survival (GRFS) post-HCT
* To determine the overall survival (OS) post-HCT
* To measure the incidence and severity of acute and chronic GVHD

Exploratory Objectives

* To measure the incidence of serious infections
* To measure the incidence and timing of engraftment
* To measure T cell immunity reconstitution parameters

ELIGIBILITY:
Inclusion Criteria:

Recipient Inclusion Criteria

a. Patients with the following diseases that are histopathologically-confirmed are eligible

* Acute myeloid, lymphoid, or mixed phenotype leukemia in complete remission (CR) or CR with incomplete hematologic recovery (CRi) or beyond first complete remission (CR1) without the presence of minimal residual disease
* Acute myeloid, leukemia, or mixed phenotype leukemia that is either:
* Not in morphologic CR with bone marrow infiltration by leukemic blasts of ≤10%, or
* In morphologic CR with evidence of minimal residual disease positivity by either multiparametric flow cytometric analysis or by a nucleic acid-based technique
* Primary refractory acute myeloid, lymphoid, or mixed phenotype leukemia
* Chronic myelogenous leukemia (accelerated, blast or second chronic phase)
* Myelodysplastic syndromes
* Myeloproliferative syndromes b. Match to the patient as follows: a. For Arm A1 (CLOSED):

  * Availability of a 8/8 or 7/8 HLA-matched donor (related or unrelated) defined by Class I (HLA-A, -B, -C) serologic typing (or higher resolution) and Class II (HLA-DRB1) molecular typing.
  * If the donor is a 7/8 HLA-match, the mismatch must be a permissive allelic mismatch as assessed by an independent HLA and transplantation expert. b. For Arm A1 and Arm A3:
  * Availability of a 8/8 HLA-matched donor (related or unrelated) defined by Class I (HLA-A, -B, -C) serologic typing (or higher resolution) and Class II (HLA-DRB1) molecular typing.

    c. For Arm B (CLOSED):
  * Availability of a haploidentical donor who is a ≥ 4/8 but <7/8 match at HLA-A, -B, -C, and -DRB1 (typed using DNA-based high-resolution methods), with at most one mismatch per locus d. For Arm C1 (CLOSED) and C2:
  * Availability of a 8/8 HLA matched donor (related or unrelated) defined by Class I (HLA-A, B, C) serologic typing (or higher resolution) and Class II (HLA DRB1) molecular typing.

    c. Age ≥ 18 and ≤75 years old at the time of enrollment. d. Left ventricular ejection fraction (LVEF) ≥ 45% e. Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50% f. Calculated creatinine clearance ≥ 50 mL/min or creatinine < 2.0 mg/dL g. SGPT and SGOT ≤ 3 x ULN, unless elevated secondary to disease Total bilirubin ≤ 2 x ULN (patients with Gilbert's syndrome may be included at the discretion of the PI or where hemolysis has been excluded h. Negative serum or urine beta-HCG test in females of childbearing potential within 3 weeks of registration i. Karnofsky performance status ≥ 70%

Donor Inclusion Criteria

1. Age ≥ 18 and ≤ 75 years of age
2. Karnofsky performance status of ≥ 70% defined by institutional standards
3. Seronegative for HIV-1 RNA PCR; HIV 1 and HIV 2 ab (antibody); HTLV-1 and HTLV-2 ab; PCR+ or sAg (surface antigen) hepatitis B ; or PCR or sAg negative for hepatitis C; negative for the Treponema palladum antibody Syphillis screen; and negative for HIV-1 and hepatitis C by nucleic acid testing (NAT) within 30 days of apheresis collection.
4. In the case that T palladum antibody tests are positive, donors must:

Be evaluated and show no evidence of syphilis infection of any stage by physical exam and history, or Have completed effective antibiotic therapy to treat syphilis, or Have a documented negative non-treponemal test (such as RPR) or in the case of a positive non-treponemal test must be evaluated by an infectious disease expert to evaluate for alternative causes of test positivity and confirm no evidence of active syphilitic disease e. Match to the patient as follows:

1. Arm A1(CLOSED):

   • Must be a related or unrelated, 8/8 or 7/8-HLA match to recipient at HLAA, -B, -C, and -DRB1. If 7/8 HLA-matched, must be with permissive allelic HLA mismatch as assessed by an independent HLA and transplantation expert.
2. Arm A2 and Arm A3:

   • Must be a related or unrelated, 8/8 HLA match to recipient at HLA A, B, C, and DRB1
3. Arm B (CLOSED):

   * Must be a haploidentical donor who is ≥ 4/8 but < 7/8 match at HLA-A, -B, -C, and -DRB1, with at most one mismatch per locus.
4. Arm C1 (CLOSED) and Arm C2:

   * Must be a related or unrelated 7/8 HLA matched to recipient at HLA A, B, C, DRB1 or -DQB1

f. Must be willing to donate PBSC for up two consecutive days g. Female donors of child-bearing potential must have a negative serum or urine beta HCG test within 3 weeks of mobilization h. Capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate i. Agreeable to 2nd donation of PBPC (or bone marrow harvest) in the event of graft failure j. The donor or legal guardian greater than 18 years of age, capable of signing an IRB approved consent form. k. Meets other criteria for donation as specified by standard NMDP guidelines (NMDP donors) or institutional standards (non-NMDP donors) l. Donors not meeting federal eligibility criterion, may nonetheless be included if either apply as follows per 21 CFR § 1271.65:

* The donor is a first-degree or second-degree blood relative of the recipient, or
* Documented urgent medical need (DUMN), meaning no comparable human cell product is available and the recipient is likely to suffer death or serious morbidity without the human cell product, as attested by the Investigator or sub-investigator

Exclusion Criteria:

Recipient Exclusion Criteria

1. Seropositive for any of the following:

   HIV antibodies; hepatitis B surface antigen (sAg); hepatitis C antibodies
2. Patients deemed candidates for fully myeloablative preparative conditioning regimens

d. Candidate for autologous transplant e. Hepatitis B or C with SGPT or SGOT > 3 x ULN f. HIV-positive g. Active uncontrolled bacterial, viral or fungal infection, defined as currently taking antimicrobial therapy and progression of clinical symptoms. h. Uncontrolled CNS disease involvement i. Pregnant or a lactating female j. Positive serum or urine beta-HCG test in females of childbearing potential within 3 weeks of registration k. Psychosocial circumstances that preclude the patient being able to go through transplant or participate responsibly in follow-up care l. Known allergy or hypersensitivity to, or intolerance of, tacrolimus m. Positive anti-donor HLA antibodies against a mismatched allele in the selected donor determined by either:

* A positive crossmatch of any titer; or
* The presence of anti-donor HLA antibody to any HLA locus n. Any uncontrolled autoimmune disease requiring active immunosuppressive treatment o. Concurrent malignancies or active disease within 1 year, except nonmelanomatous skin cancers that have been curatively resected

Donor Exclusion Criteria

1. Evidence of active infection
2. Seropositive for HIV-1 or-2, HTLV-1 or -2
3. Medical, physical, or psychological reason that would place the donor at increased risk for complications from growth factor or leukapheresis
4. Lactating female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Determine the GVHD-free relapse-free survival (GRFS) post-HCT ( Arm-A) | 12 months
  Clinical effect will be assessed as graft vs host disease (GVHD)-free relapse free survival (GRFS), GVHD-free is defined as no GVHD symptoms, and relapse free survival is defined as survival at 12 months without relapse. The outcome will be measured in Arm A only.
Determine the overall survival (OS) post-HCT ( Arm-B) | 2 years
  Overall survival is measured as number of participants alive. Alive at the time of last observation will be censored.
Incidence of Grade III-IV acute GVHD | At baseline, day +30, 60, 90, 180, year 1 and year 2
  Acute GVHD will be staged and graded per Mount Sinai Acute GvHD International Consortium (MAGIC) Standardization criteria.
The incidence and timing of primary graft failure | 2 years from the Day 0 (day of CD34+ peripheral blood stem cell infusion
  Primary graft failure is defined as being alive with donor CD3 chimerism <5% at day +30 after transplant without recovery of neutrophils (i.e. without achieving an absolute neutrophil count [ANC] ≥ 500/mm3 for 3 consecutive days) at Day+28
Donor CD3 chimerism at Day+60 post-HCT | 2 years from the Day 0 (day of CD34+ peripheral blood stem cell infusion)
  Defined as a percentage on donor CD3 cells chimerism at day +60 after transplantation.

SECONDARY OUTCOMES:
GVHD-relapse-free survival | 12 months
  Clinical effect will be assessed as graft vs host disease (GVHD)-free relapse free survival (GRFS), GVHD-free is defined as no GVHD grade 3 and 4, and relapse free survival is defined as survival at 12 months without relapse.
Overall survival | 12 months
  Overall survival is measured as number of participants alive. Alive at the time of last observation will be censored.
Secondary graft failure | from Day 0 through 100 days
  Secondary graft failure (defined by donor CD3 chimerism <5% at day +30 after transplant) and neutrophil engraftment followed by subsequent decline in ANC < 500/mm3 unresponsive to growth factor therapy, by Day +100
Treatment-emergent adverse events (TEAs) | from Day 0 through 100 days
  TEAEs will be categorized by the System Organ Class and preferred term and will be graded according to the CTCAE version 5.0
Acute GVHD (all grades) | from Day 0 through 100 days
  Acute GVHD (all grades) will be reported
Steroid-refractory acute GVHD | within 3-5 days of therapy onset
  Steroid refractory acute GVHD will be defined as per the EBMT-NIH-CIBMTR Task Force position statement
Non-relapse mortality (NRM) | 12 months
  Non-relapse mortality is measured as number of participants died without relapse/ recurrent disease. Subjects without evidence of relapse/progression at last follow-up date or date of death will be censored.
Disease-free survival (DFS) | 12 months
  Overall survival is measured as number of participants alive and in remission. Alive in remission at the time of last observation will be censored.
Chronic GVHD (limited or extensive) | from Day 0 through Year 2
  Chronic GVHD will be diagnosed per 2014 International NIH Chronic GVHD Diagnosis and Staging Consensus Working Group criteria (Jagasia 2015). Chronic GVHD scored according to the first day of chronic GVHD onset will be used to calculate cumulative incidence curves. Subjects will be followed for 2 years from the Day 0 (day of CD34+ peripheral blood stem cell infusion) for estimation of cGVHD incidence.

OTHER OUTCOMES:
Time to Neutrophil engraftment | from Day 0 through 100 days
  Neutrophil engraftment is defined as having an ANC ≥ 500 cells/µL for three consecutive days. The first of three days will be designated as the day of engraftment.
Time to Platelet engraftment | from Day 0 through 100 days
  Platelet engraftment is defined as achieving a platelet count > 20,000 cells/µL for three consecutive days without platelet transfusion in the preceding 7 days. The first of three days will be designated as the day of engraftment.
Incidence of serious infections (grade 2 and greater) | from Day 0 through 100 days
  Incidence of serious infections will be measured as event of infections that led to hospitalization or death or required antibiotic treatment. Infections will be graded according to the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Everett Meyer, MD,PhD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No